CLINICAL TRIAL: NCT04678752
Title: PATHWEIGH: Pragmatic Weight Management in Primary Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-1954; 1R18DK127003 (NIH)
Record Dates: First submitted 2020-11-24; First posted 2020-12-22 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-04

CONDITIONS: Obesity
Keywords: Obesity; Primary Care; Electronic Health Record
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Effectiveness-Implementation Hybrid Type 1 Study using a Stepped Wedge Cluster Randomized Trial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Each primary care provider will administer weight loss care per their standard practice.
  Interventions: Other: Control
- PATHWEIGH (Experimental): A weight management care path that support primary care both through the EHR and training for the clinicians.
  Interventions: Other: Weight management care path

INTERVENTIONS:
Other: Weight management care path — * Documentation and data capture built in the Electronic Health Record
  * Clinical data support that suggests weight loss approach(es)
  * Tracking of weight loss progress and weight loss maintenance during patient visits to guide the patient-clinician conversation
  * Diagnosis and billing in EHR automatically adds the diagnosis of overweight or obesity and links the most common weight-related co-morbidities to ensure adequate provider reimbursement
  * Evidence-based online training on weight management for clinicians
  * Practice quality improvement and training for use of PATHWEIGH for weight-prioritized visits through practice coaches/facilitators
  * Consultation support by practice facilitators with implementing PATHWEIGH and by obesity providers for clinicians with creating patient treatment plans
  Arms: PATHWEIGH
Other: Control — Within primary care the option to select "Obesity brief HPI", this is a brief historical intake of a patient's weight - when either they or their clinician decides to have a weight-prioritized visit. It is intended to initiate a discussion regarding potential strategies for weight loss (often "eat less, exercise more"). The provider has the discretion to augment or add support as they see fit.
  Arms: Standard of Care

SUMMARY:
The study examines patient weight loss and maintenance, associated predictors (patient health characteristics and demographics), and contextual factors in the practice environment that influence the intervention's adoption, implementation, and sustainability. This will be achieved through a mixed methods implementation study including collection and analysis of de-identified clinical data, surveys, observations, and interviews.

DETAILED DESCRIPTION:
This study will investigate how PATHWEIGH, a weight management tool built into the EPIC electronic health record, in combination with clinician and staff training on the use of PATHWEIGH as a tool, education on effective weight management practices, and practice facilitation to support implementation can facilitate weight loss and maintenance for primary care patients. The study examines patient weight loss and maintenance, associated predictors (patient health characteristics and demographics), and contextual factors in the practice environment that influence the intervention's adoption, implementation, and sustainability. This will be achieved through a mixed methods implementation study including collection and analysis of de-identified clinical data, surveys, observations, and interviews.

This study is being conducted because despite obesity being the leading cause of preventable death in the U.S. and a major risk factor for disease, people with any degree of overweight or obesity are rarely offered anything other than lifestyle advice, rather than more rigorous and evidence-based weight management strategies. Poor reimbursement for weight-related visits, competing priorities, lack of appropriate tools, and limited time in visits also prevent more widespread use of weight management interventions. PATHWEIGH helps primary care clinicians and teams prioritize weight management with their patients when appropriate and ensures that they have the tools and knowledge handy to do so effectively. As part of the assessment of the PATHWEIGH intervention, the study will identify predictors of patient weight loss and weight loss maintenance using mediator and moderator analysis. Relevant factors (patient demographics, health metrics (e.g. vital signs, anthropometrics, comorbidities), behaviors and goals, provider age, sex, years and % time practicing, and clinic information (e.g. size, location, culture scale)) will be evaluated by including interaction terms between the treatment variable and possible moderating variables in outcome regression models .

ELIGIBILITY:
Clinician Inclusion Criteria:

* Affiliated with a participating primary care practice
* Provide care for adult patients (>=18 years old)

Patient Inclusion Criteria:

* All adult patients (age >18 years)
* BMI >25 kg/m2
* Appointment at a primary care clinic participating in the study

Patient Exclusion Criteria:

* Unable to participate in weight loss treatment due to factors such as cognitive deficits, non-home residence, or limited life expectancy.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2020-03-17 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Patient weight trajectories over the 6 months after the initial weight measured in the usual care and intervention phases | 0 to 6 months
  Change in patient weight trajectories 0-6 months after the initial weight measurement in the usual care and intervention phases.
Patient weight maintenance, as measured by patient weight trajectories from 6 to 18 months after the initial weight measurement, in the usual care and intervention phases | 6 to 18 months
  Change in patient weight trajectories from 6 to 18 months after the initial weight measurement in the usual care and intervention phases.

SECONDARY OUTCOMES:
Patient weight maintenance, as measured by patient weight trajectories from 6 to 18 months after the initial weight measurement, in the usual care and intervention phases stratified by those received vs. did not receive discernible weight-related care | 6 to 18 months
  Change in weight from 6 to 18 months after the initial weight measurement in the usual care and intervention phases stratified by those who did and did not receive discernible weight related care.

OTHER OUTCOMES:
Reach - The representativeness of individuals who participate in the trial. | Baseline and each 1 year step after
  Individual participants enrolled on the trial versus the number of patients eligible for the trial will be assessed within the electronic medical record.
Qualitative assessment of the reach of patient recruitment | 6 months post intervention start
  Interviews with a purposefully selected sample of patients to measure factors that impact patient recruitment to the study.
Adoption - The representativeness of providers who initiate the intervention | Baseline and at each 1 year step
  The proportion of medical providers who provide the PATHWEIGH intervention to patients over medical providers who were eligible but chose not to provide the PATHWEIGH intervention will be calculated overall and within each participating clinic.
Qualitative assessment of adoption of the intervention by medical providers. | 1 year post intervention start/cohort
  Qualitative interviews of a purposefully selected sample of providers will be conducted to understand reasons and barriers to adoption of PATHWEIGH.
Implementation - The intervention agents' fidelity to the various elements of the intervention's protocol including consistency of delivery as intended and the time and cost of the intervention | Every 6 months for 5 years
  The number of medical providers who provided the PATHWEIGH intervention to patients correctly (meeting fidelity criteria) which will be abstracted from the medical record.
Implementation - The intervention agents' fidelity to the various elements of the intervention's protocol including consistency of delivery as intended and the time and cost of the intervention | 6 months post intervention for each cohort through study end
  Interviews with a purposefully selected sample of providers will be conducted to measure factors that impact the implementation of PATHWEIGH.
Maintenance - The proportion of patients that maintained weight loss at 18 months post enrollment. | 18 months post enrollment
  Patients will be weighed and the difference from initial weight-prioritized visit.
Maintenance - The extent to which the intervention becomes part of practice | 1 year post intervention start cohort up till year 5 of the study
  Each practice will be evaluated for the extent to which they continue to use the PATHWEIGH intervention via medical record review indicating intervention use amongst eligible patients.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Perreault, MD, Principal Investigator — University of Colorado, Denver; Jodi S Holtrop, PhD, Principal Investigator — University of Colorado, Denver
Locations (64):
- United States (64):
  - UCHealth Primary Care - Arvada West, Arvada, Colorado
  - UCHealth Primary Care - Quincy, Aurora, Colorado
  - UCHealth Executive Health Services - Anschutz Medical Campus, Aurora, Colorado
  - UCHealth Internal Medicine - Anschutz Medical Campus, Aurora, Colorado
  - UCHealth Seniors Clinic - Anschutz Medical Campus, Aurora, Colorado
  - UCHealth Women's Integrated Services in Health - Anschutz Medical Campus, Aurora, Colorado
  - UCHealth Family Medicine - Boulder, Boulder, Colorado
  - UCHealth CU Family Medicine - Depot Hill, Broomfield, Colorado
  - UCHealth Primary Care - Broomfield, Broomfield, Colorado
  - UCHealth Primary Care - Castle Rock, Castle Rock, Colorado
  - UCHealth CU Family Medicine - Centennial, Centennial, Colorado
  - UCHealth Primary Care and Sports Medicine Clinic - Lake Plaza, Colorado Springs, Colorado
  - UCHealth Primary Care - Fontanero, Colorado Springs, Colorado
  - UCHealth Internal Medicine - Printers Park, Colorado Springs, Colorado
  - UCHealth Sports Medicine Clinic - Printers Park, Colorado Springs, Colorado
  - UCHealth Primary Care - Academy, Colorado Springs, Colorado
  - UCHealth Primary Care - Rockrimmon, Colorado Springs, Colorado
  - UCHealth Aspen Creek Medical Center, Colorado Springs, Colorado
  - UCHealth Primary Care - Briargate, Colorado Springs, Colorado
  - UCHealth Primary Care - Chapel Hills, Colorado Springs, Colorado
  - UCHealth Primary Care - Scarborough, Colorado Springs, Colorado
  - UCHealth Primary Care - Craig, Craig, Colorado
  - UCHealth Primary Care - Cripple Creek, Cripple Creek, Colorado
  - UCHealth Primary Care - Steele Street, Denver, Colorado
  - UCHealth CU Internal Medicine - Garfield, Denver, Colorado
  - UCHealth Primary Care - Uptown, Denver, Colorado
  - UCHealth Internal Medicine - Lowry, Denver, Colorado
  - UCHealth A.F. Williams Family Medicine Clinic - Central Park, Denver, Colorado
  - UCHealth Primary Care - Estes Park, Estes Park, Colorado
  - UCHealth Primary Care - Falcon, Falcon, Colorado
  - UCHealth Family Medicine - Firestone, Firestone, Colorado
  - UCHealth Family Medicine Center - Fort Collins, Fort Collins, Colorado
  - UCHealth Internal Medicine - Prospect, Fort Collins, Colorado
  - UCHealth Internal Medicine - Snow Mesa, Fort Collins, Colorado
  - UCHealth Internal Medicine and Pediatric Care Clinic - Snow Mesa, Fort Collins, Colorado
  - UCHealth Internal Medicine - Greeley Midtown, Greeley, Colorado
  - UCHealth Family Medicine - Greeley, Greeley, Colorado
  - UCHealth Internal Medicine - Greeley, Greeley, Colorado
  - UCHealth CU Family Medicine - Landmark, Greenwood Village, Colorado
  - UCHealth Primary Care - Greenwood Village, Greenwood Village, Colorado
  - UCHealth Primary Care - Highlands Ranch, Highlands Ranch, Colorado
  - UCHealth Family Medicine - Littleton, Highlands Ranch, Colorado
  - UCHealth Primary Care - Sterling Ranch, Littleton, Colorado
  - UCHealth Primary Care - Lone Tree, Lone Tree, Colorado
  - UCHealth Primary Care - Yosemite, Lone Tree, Colorado
  - UCHealth Women's Integrated Services in Health - Lone Tree, Lone Tree, Colorado
  - UCHealth Family Medicine - Longmont, Longmont, Colorado
  - UCHealth Internal Medicine - Longmont, Longmont, Colorado
  - UCHealth Longmont Clinic, Longmont, Colorado
  - UCHealth Orchards Medical Center, Loveland, Colorado
  - UCHealth Family Medicine - North Loveland, Loveland, Colorado
  - UCHealth Internal Medicine - East Loveland, Loveland, Colorado
  - UCHealth Internal Medicine - Orchards, Loveland, Colorado
  - UCHealth Primary Care - Monument, Monument, Colorado
  - UCHealth Primary Care - Hilltop, Parker, Colorado
  - UCHealth Primary Care and Women's Wellness - Stonegate, Parker, Colorado
  - UCHealth Primary Care - Sterling, Sterling, Colorado
  - UCHealth Primary Care - Timnath, Timnath, Colorado
  - UCHealth Family Medicine - Westminster, Westminster, Colorado
  - UCHealth Family Medicine - Windsor, Windsor, Colorado
  - UCHealth Family Medicine - Woodland Park, Woodland Park, Colorado
  - Little Snake River Clinic - Managed by UCHealth Yampa Valley Medical Center, Baggs, Wyoming
  - UCHealth Cheyenne Medical Specialists, Cheyenne, Wyoming
  - UCHealth Primary Care - Cheyenne, Cheyenne, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
Data sharing from 1R18DK127003 will comply with policies from the NIH https://grants.nih.gov/grants/policy/data_sharing/), ICMJE (http://www.icmje.org/recommendations/browse/publishing-and-editorial-issues/clinical-trial-registration.html#two), as well as our IRB. No individual participant data will be shared. Data that will be publicly available (through their publication) will include study protocol, analysis plan, and results presented in aggregate. Additional information may be shared upon request.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Perreault L, Pan Q, Rodriguez C, Gritz RM, Smith PC, Kramer ES, Tolle L, Connelly L, Tietbohl C, Williams J 2nd, Holtrop JS. Implementation and effectiveness of a care process to prioritize weight management in primary care: a stepped-wedge cluster-randomized trial. Nat Med. 2025 Dec 11. doi: 10.1038/s41591-025-04051-5. Online ahead of print. PMID 41381746
- [Derived] Perreault L, Suresh K, Rodriguez C, Dickinson LM, Willems E, Smith PC, Williams J Jr, Gritz RM, Holtrop JS. Baseline Characteristics of PATHWEIGH: A Stepped-Wedge Cluster Randomized Study for Weight Management in Primary Care. Ann Fam Med. 2023 May-Jun;21(3):249-255. doi: 10.1370/afm.2966. PMID 37217322
- [Derived] Suresh K, Holtrop JS, Dickinson LM, Willems E, Smith PC, Gritz RM, Perreault L. PATHWEIGH, pragmatic weight management in adult patients in primary care in Colorado, USA: study protocol for a stepped wedge cluster randomized trial. Trials. 2022 Jan 10;23(1):26. doi: 10.1186/s13063-021-05954-7. PMID 35012628